CLINICAL TRIAL: NCT00802295
Title: Influence of Ovarian Stimulation and Embryo Aneuploidy
Brief Title: Aneuploidies and Different Stimulation Protocols
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Jose Remohi Jimenez, IVI Valencia
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: VLC-JR-0204-307-11
Record Dates: First submitted 2008-12-03; First posted 2008-12-04 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Aneuploidy
Keywords: Ovarian; hyperstimulation; Embryo; Aneuploidy; Ovarian hyperstimulation and Embryo Aneuploidy Rates
MeSH Terms: conditions — Aneuploidy | interventions — Gonadotropins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard dosis protocol (Active Comparator): Administration of standard dosis of gonadotrophins for ovarian stimulation.
  Interventions: Drug: Gonadotrophins
- 2 (Experimental): Administration of low dosis of Gonadotrophins for ovarian stimulation
  Interventions: Drug: Low dosis Gonadotrophin

INTERVENTIONS:
Drug: Gonadotrophins — Administration of standard ovarian stimulation protocol
  Arms: standard dosis protocol
Drug: Low dosis Gonadotrophin
  Arms: 2

SUMMARY:
Our working hypothesis is that patients undergoing "in vitro" fertilization (IVF) with higher response to ovarian stimulation protocols recover a higher number of oocytes and, this elevated response could be translated into increased incidence of chromosomally abnormal embryos. Our objective is to develop a prospective study on healthy young donors, with a previous cycle with high ovarian response (>20 oocytes and/or E2 levels the day of the hCG injection >3000 pg/mL), but without developing mild or severe hyperstimulation syndrome. After signing a proper written consent, these donors would agree to undergo two subsequent stimulation cycles following two different protocols. In one cycle the stimulation pattern would be similar to the previous one, with elevated response and, in another cycle the amount of gonadotropins would be cut down in order to obtain lower ovarian response. Oocytes obtained in each cycle would be donated to anonymous recipients and after fertilization, embryo quality and chromosomal status of the resulting embryos would be evaluated. Preimplantation genetic diagnosis (PGD) will be performed on day-3 embryos and chromosomes 13, 15, 16, 17, 18, 21, 22, X and Y would be analyzed by fluorescence "in situ" hybridization (FISH).

ELIGIBILITY:
Inclusion Criteria:

* Healthy women between 18 - 29
* with previous cycle with standard dosis of Gonadotrophin and high response to the treatment (> 20 oocytes)
* No symptom of OHSS

Exclusion Criteria:

* donors with 2 previous miscarriages
* PCO
* Severe Male Factor

Ages: 18 Years to 29 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Aneuploidy rate with two different stimulation protocols. | three months

SECONDARY OUTCOMES:
Normal blastocyst rate | three months

CONTACTS AND LOCATIONS:
Overall Officials: Jose Remohi, MD PhD, Principal Investigator — IVI Valencia
Locations (1):
- Instituto Valenciano de Infertilidad, Valencia, Spain

REFERENCES:
- [Derived] Rubio C, Mercader A, Alama P, Lizan C, Rodrigo L, Labarta E, Melo M, Pellicer A, Remohi J. Prospective cohort study in high responder oocyte donors using two hormonal stimulation protocols: impact on embryo aneuploidy and development. Hum Reprod. 2010 Sep;25(9):2290-7. doi: 10.1093/humrep/deq174. Epub 2010 Jul 13. PMID 20627979